CLINICAL TRIAL: NCT07211126
Title: The Real-World Control-IQ Glycemic Control and Quality of Life Study in Type 1 Diabetes in France
Acronym: RECORD-IQ
Status: Not yet recruiting | Type: Observational
Sponsor: Tandem Diabetes Care, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TP-0018999
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Control-IQ; t:slim X2 insulin pump; Control-IQ technology; DKA; severe hypoglycemia; automated insulin dosing; automated insulin delivery; quality of life; type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Control-IQ System: Participants will use the Control-IQ System as per standard of care.
  Interventions: Device: t:slim X2 insulin pump with Control-IQ technology (Control-IQ System)

INTERVENTIONS:
Device: t:slim X2 insulin pump with Control-IQ technology (Control-IQ System) — Participants enrolled in the study will start use of the t:slim X2 insulin pump with Control-IQ technology (Control-IQ System) with Dexcom G6 or Dexcom G7, and be followed for 12 months.

SUMMARY:
This post-market surveillance study is primarily designed to demonstrate the ongoing safety of the Control-IQ system, the ongoing performance of glycemic control and quality of life with Control-IQ system use, and the rate of use of the Control-IQ system. The system will be assessed in all approved populations during the first 12 months of use.

DETAILED DESCRIPTION:
This post-market surveillance study is a single-arm, prospective cohort study. It is designed to:

1. Demonstrate, in the post-approval setting, the safety of the Control-IQ System for the management of type 1 diabetes by assessing the rate of severe metabolic complications (severe hypoglycemia and/or diabetic ketoacidosis).
2. Determine glycemic outcomes during real-world use of the Control-IQ System over 12 months post-initiation.
3. Demonstrate patient-reported satisfaction with the device, trust in the Control-IQ System, usability of the system, and improved quality of life.
4. Describe the real-world use of the Control-IQ System.

ELIGIBILITY:
Inclusion Criteria:

* Clinician-confirmed type 1 diabetes and for whom the site has initiated the t:slim X2 insulin pump with Control-IQ technology (Control-IQ System) with a Dexcom G6 or G7 CGM sensor.
* Age ≥ 6 years at enrollment.
* Using an insulin approved for use in the pump.
* Ability for patient or parent/guardian to respond to alerts and alarms, and to provide basic diabetes self-management.
* Reside full-time in mainland France.
* Have an email address and mobile phone number
* Participant or participant's parent/guardian has read and understood the information notice and has agreed to participate in the study. This includes agreeing to :

  1. use Control-IQ technology, and to continue use for at least 12 consecutive months after study enrollment.
  2. the reuse of their clinical data including HbA1c results, obtained at most 4 months prior to enrollment, and as available according to the standard of care during the next 12 months.
  3. complete questionnaires per the study protocol.

Exclusion Criteria:

* A medical or other condition, or medications being taken that, in the investigator's judgement would be a safety concern for participation in the study.
* Patients considered vulnerable under French law.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All individuals with Type 1 Diabetes age 6+, who start therapy with the t:slim X2 insulin pump with Control-IQ technology (Control-IQ System) with a Dexcom G6 or Dexcom G7 and meet eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Rate of diabetic ketoacidosis (DKA). | 12 months
  The incidence rate of diabetic ketoacidosis (DKA) will be calculated by dividing the total number of events observed in the entire cohort over the 12-month follow-up period. Results will be expressed as the number of events per 100 patient-years.
Rate of severe hypoglycemia (SH) | 12 months
  The incidence rate of severe hypoglycemia (SH) will be calculated by dividing the total number of events observed in the entire cohort over the 12-month follow-up period. Results will be expressed as the number of events per 100 patient-years.

SECONDARY OUTCOMES:
Time in Range 70-180 mg/dL (TIR) | 12 months
  The change in (%) time spent within range, defined as the proportion of sensor glucose concentration within the target range of 70-180 mg/dL, between baseline and 12 months.
Time above 180 mg/dL | 12 months
  The change in (%) time spent above 180 mg/dL, defined as the proportion of sensor glucose concentration above 180 mg/dL, between baseline and 12 months.
Time above 250 mg/dL | 12 months
  The change in (%) time spent above 250 mg/dL, defined as the proportion of sensor glucose concentration above 250 mg/dL, between baseline and 12 months.
Time less than 70 mg/dL | 12 months
  The change in (%) time spent less than 70 mg/dL, defined as the proportion of sensor glucose concentration less than 70 mg/dL, between baseline and 12 months.
Time less than 54 mg/dL | 12 months
  The change in (%) time spent less than 54 mg/dL, defined as the proportion of sensor glucose concentration less than 54 mg/dL, between baseline and 12 months.
Treatment Satisfaction | 12 months
  To evaluate treatment satisfaction based on the Diabetes Treatment Satisfaction Questionnaire status (DTSQs) scores at baseline through 12 months.
System Usability | 12 months
  To evaluate treatment satisfaction based on the System Usability Scale (SUS) scores at baseline through 12 months.
Quality of Life Change | 12 months
  To evaluate change in quality of life based on the EQ-5D scores at baseline through 12 months.
Fear of Hypoglycemic Events Change | 12 months
  To evaluate change in fear of hypoglycemic events based on the Hypoglycemia Fear Survey (HFS) from baseline through 12 months.
Rate of use of the system | 12 months
  To determine the rate of use of the system as established by % time in closed-loop, from baseline through 12 months.

IPD SHARING:
Plan to Share IPD: No